CLINICAL TRIAL: NCT07056582
Title: Pre-emptive Analgesia Using Nebulized Ketamine Versus Nebulized Dexmedetomidine in Endoscopic Nasal Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Thabet Abdelhameed, Resident , Anesthesia , Surgical Icu , Pain management Faculty of Medicine Sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Soh-Med--25-4-08MS
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Nose Diseases
MeSH Terms: conditions — Nose Diseases | interventions — Dexmedetomidine; Ketamine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group D : will receive dexmedetomidine (Active Comparator): Patients will receive nebulized dexmedetomidine 50 μg (0.5 ml +normal saline 0.9% up to 3 ml) 15 minutes prior to the onset of surgery.
  Interventions: Drug: Dexmedetomidine
- group K : will receive ketamine (Active Comparator): patients will receive nebulized ketamine 50 mg (1 ml + normal saline 0.9%up to 3 ml) 15 minutes prior to the onset of surgery.
  Interventions: Drug: Ketamine
- group C: will receive .9% saline (Placebo Comparator): Patients will receive nebulized normal saline 0.9% (3 ml) 15 minutes prior to the onset of surgery.
  Interventions: Drug: 0.9%sodium chloride

INTERVENTIONS:
Drug: Dexmedetomidine — patients in this group will receive nebulized Dexmedetomidine before onset of surgery
  Arms: group D : will receive dexmedetomidine
Drug: Ketamine — patients in this group will receive nebulized ketamine before onset of surgery
  Arms: group K : will receive ketamine
Drug: 0.9%sodium chloride — patients in this group will receive nebulized 0.9% normal saline before onset of surgery
  Arms: group C: will receive .9% saline

SUMMARY:
this study aims to compare the efficacy of pre-emptive nebulized ketamine versus nebulized dexmedetomidine for post operative pain relief in endoscopic nasal surgery

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 20 and 60,
* both sexes,
* American Society of Anesthesiologists physical status I to II
* BMI ≥18≤30 kg/m²

Exclusion Criteria:

* Patient refusal.
* patients with advanced respiratory, renal, hepatic, neurological, or psychiatric disease, pregnant or nursing women.
* patients with a history of allergies to any study drugs.
* patients who had used central nervous system depressants or analgesics within the previous 24 hours.
* patients with hypertension, hypotension, or bradycardia.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
This study aims to assess the efficacy of nebulized dexmedetomidine vs nebulized ketamine to achieve good postoperative pain management in patients undergoing endoscopic nasal surgeries. | 24 hours after operation
  post operative pain management by VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Result] Parthasarathy S, Krishnapriyanka KJ, Saravanan B. Effectiveness of pre-emptive nerve block on opioid consumption in patients undergoing nasal surgery under general anaesthesia: A double-blinded randomised controlled study. Indian J Anaesth. 2022 Feb;66(2):133-139. doi: 10.4103/ija.ija_813_21. Epub 2022 Feb 24. PMID 35359478
- [Result] Prasant NVSN, Mohapatro S, Jena J, Moda N. Comparison of Preoperative Nebulization with 4% Lignocaine and Ketamine in Reduction of Incidence of Postoperative Sore Throat. Anesth Essays Res. 2021 Jul-Sep;15(3):316-320. doi: 10.4103/aer.aer_105_21. Epub 2022 Feb 14. PMID 35320968
- [Result] Cai Y, Xu H, Yan J, Zhang L, Lu Y. Molecular targets and mechanism of action of dexmedetomidine in treatment of ischemia/reperfusion injury. Mol Med Rep. 2014 May;9(5):1542-50. doi: 10.3892/mmr.2014.2034. Epub 2014 Mar 10. PMID 24627001